CLINICAL TRIAL: NCT01245049
Title: Immunogenicity and Safety of GSK Biologicals' dTpa-IPV Vaccine (Boostrix Polio) as a Booster Dose in 3 and 4-year-old Children
Brief Title: Immunogenicity and Safety of GSK Biologicals' Boostrix Polio Vaccine in 3 and 4-year-old Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111763
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-06

CONDITIONS: Acellular Pertussis; Poliomyelitis; Tetanus; Diphtheria
Keywords: MMR; dTpa-IPV; Boostrix Polio; Repevax; Priorix
MeSH Terms: conditions — Poliomyelitis; Tetanus; Diphtheria

ARMS (2):
- BOOSTRIX POLIO GROUP (Experimental): Healthy male or female children of 3 or 4 years of age, who were previously vaccinated with 3 doses of Infanrix™ and Polio™ vaccines in the German household contact study (APV-039), additionally received 1 booster dose of Boostrix™ Polio vaccine co-administered with Priorix™ vaccine at Day 0. Boostrix™ Polio vaccine was administered intramuscularly in the deltoid muscle of the left arm, while Priorix™ vaccine was administered subcutaneously in the deltoid region of the right arm or as an intramuscular injection into the deltoid muscle of the right arm.
  Interventions: Biological: Boostrix PolioTM; Biological: PriorixTM
- REPEVAX GROUP (Active Comparator): Healthy male or female children of 3 or 4 years of age, who were previously vaccinated with 3 doses of Infanrix™ and Polio™ vaccines in the German household contact study (APV-039), additionally received 1 booster dose of Repevax™ vaccine co-administered with Priorix™ vaccine at Day 0. Repevax™ vaccine was administered intramuscularly in the deltoid muscle of the arm, while Priorix™ vaccine was administered subcutaneously in the deltoid region of the right arn or as an intramuscular injection into the deltoid muscle of the right arm.
  Interventions: Biological: RepevaxTM; Biological: PriorixTM

INTERVENTIONS:
Biological: Boostrix PolioTM — Single dose, intramuscular administration.
  Arms: BOOSTRIX POLIO GROUP
Biological: RepevaxTM — Single dose, intramuscular administration.
  Arms: REPEVAX GROUP
Biological: PriorixTM — Single dose, intramuscular or subcutaneous administration.

SUMMARY:
The purpose of the study is to compare the immunogenicity and safety of a booster dose of BoostrixTM Polio to that of Sanofi Pasteur MSD's RepevaxTM, when co-administered with a second dose of PriorixTM, in healthy 3 and 4-year-old children.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female child of 3 or 4 years of age at the time of booster vaccination (up to, but excluding 5 years of age).
* Subjects who have received a complete three-dose primary vaccination with diphtheria-tetanus-acellular pertussis (DTPa) vaccine and inactivated poliovirus (IPV) vaccine in the first six months of life, in line with recommendations in the United Kingdom (UK).
* Subjects who received a first dose of a live attenuated measles-mumps-rubella vaccine within the second year of life, in line with recommendations in the UK.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject at the time of enrolment.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period, with the exception of inactivated influenza vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous booster vaccination against diphtheria, tetanus, pertussis, poliomyelitis since primary vaccination in the first year of life.
* Previous measles, mumps and/or rubella second dose vaccination.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, poliomyelitis, measles, mumps and/or rubella disease.
* Known exposure to measles, mumps and/or rubella within 30 days prior to study start.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulin and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation.
* Occurrence of any of the following adverse events after a previous administration of a DTP vaccine:

  * Hypersensitivity reaction to any component of the vaccine;
  * Encephalopathy of unknown aetiology occurring within 7 days following previous vaccination with pertussis-containing vaccine;
  * Fever >= 40°C within 48 hours of vaccination, not due to another identifiable cause;
  * Collapse or shock-like state within 48 hours of vaccination;
  * Convulsions with or without fever, occurring within 3 days of vaccination.
* Acute disease and/or fever at the time of enrolment or within 24 hours of study vaccine administration.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 387 (Actual)
Dates: Start 2011-04-01; Primary Completion 2012-03-27 (Actual); Study Completion 2012-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United Kingdom (13):
  - GSK Investigational Site, St Austell, Cornwall
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Axbridge, Somerset
  - GSK Investigational Site, Taunton, Somerset
  - GSK Investigational Site, Atherstone, Warwickshire
  - GSK Investigational Site, Bangor
  - GSK Investigational Site, Bolton, Nr Manchester
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Crumpsall, Manchester
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Lancashire
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Randalstown

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Marlow R, Kuriyakose S, Mesaros N, Han HH, Tomlinson R, Faust SN, Snape MD, Pollard AJ, Finn A. A phase III, open-label, randomised multicentre study to evaluate the immunogenicity and safety of a booster dose of two different reduced antigen diphtheria-tetanus-acellular pertussis-polio vaccines, when co-administered with measles-mumps-rubella vaccine in 3 and 4-year-old healthy children in the UK. Vaccine. 2018 Apr 19;36(17):2300-2306. doi: 10.1016/j.vaccine.2018.03.021. Epub 2018 Mar 22. PMID 29576304
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 subjects did not receive vaccination.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Boostrix Polio Group: Healthy male or female children of 3 or 4 years of age, who were previously vaccinated with 3 doses of Infanrix and Polio vaccines in the German household contact study (APV-039), additionally received 1 booster dose of Boostrix Polio vaccine co-administered with Priorix vaccine at Day 0. Boostrix Polio vaccine was administered intramuscularly in the deltoid muscle of the left arm, while Priorix vaccine was administered subcutaneously in the deltoid region of the right arm or as an intramuscular injection into the deltoid muscle of the right arm.
- Repevax Group: Healthy male or female children of 3 or 4 years of age, who were previously vaccinated with 3 doses of Infanrix and Polio vaccines in the German household contact study (APV-039), additionally received 1 booster dose of Repevax vaccine co-administered with Priorix vaccine at Day 0. Repevax vaccine was administered intramuscularly in the deltoid muscle of the arm, while Priorix vaccine was administered subcutaneously in the deltoid region of the right arn or as an intramuscular injection into the deltoid muscle of the right arm.
Period: Overall Study
Arm/Group | Boostrix Polio Group | Repevax Group
Started | 255 | 130
Completed | 254 | 126
Not Completed | 1 | 4
Not completed — Migrated/moved from study area | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix Polio Group | Repevax Group | Total
Number analyzed (Participants) | 255 | 130 | 385
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.1 (0.2) | 3.1 (0.2) | 3.1 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 65 | 188
  Male | 132 | 65 | 197
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 2 | 4 | 6
  Asian-Central/South Asian heritage | 4 | 4 | 8
  Asian-South East Asian heritage | 3 | 1 | 4
  White-Arabic/North African heritage | 2 | 1 | 3
  White-Caucasian/European heritage | 226 | 111 | 337
  Not specified | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Booster Response to Diphtheria (D) and Tetanus (T) Antigens
Description: Booster response was defined as: For initially seronegative subjects [i.e. pre-vaccination concentration below (<) cut-off value of 0.1 international units per milliliter (IU/mL)] antibody concentrations at least four times the assay cut-off [post vaccination concentration greater than or equal to (≥) 0.4 IU/ml]. For initially seropositive subjects (pre-vaccination concentration ≥ 0.1 IU/ml), an increase in antibody concentrations of at least four times the Pre booster vaccination concentration.
Time Frame: At Month 1, one month after the booster vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 177 | 90
Participants
  Anti-D | 176 | 90
  Anti-T: number analyzed (Participants) | 176 | 90
  Anti-T | 173 | 90
Statistical Analysis 1: Comparison: Boostrix Polio Group vs Repevax Group; Non-inferiority in terms of booster response to D; Test type: Non-Inferiority — To assess the Non-inferiority of the Boostrix Polio Group compared to the Repevax Group in terms of booster response to diphtheria, standardized asymptotic 95% CI for the groups'difference [Repevax Group minus Boostrix Polio Group] was computed. Non-inferiority criterion: Upper limit of the 95% CI of the groups' difference in booster response rate ≤10%; Standardized asymptotic; Percentage difference = 0.56, 95% CI 2-sided [-3.55 to 3.14]
Statistical Analysis 2: Comparison: Boostrix Polio Group vs Repevax Group; Non-inferiority in terms of booster response to T; Test type: Non-Inferiority — To assess the Non-inferiority of the Boostrix Polio Group compared to the Repevax Group in terms of booster response to tetanus, standardized asymptotic 95% CI for the groups' difference [Repevax Group minus Boostrix Polio Group] was computed. Non-inferiority criterion: Upper limit of the 95% CI of the groups' difference in booster response rate ≤10%; Percentage difference = 1.7, 95% CI 2-sided [-2.43 to 4.9]

2. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 1, one month after the booster vaccination
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 195 | 96
EL.U/mL
  Anti-PT: number analyzed (Participants) | 194 | 96
  Anti-PT | 70.1 [62.2 to 79] | 47.8 [39.9 to 57.3]
  Anti-FHA: number analyzed (Participants) | 195 | 95
  Anti-FHA | 358.3 [312.5 to 410.8] | 164.8 [138.5 to 196.1]
  Anti-PRN: number analyzed (Participants) | 195 | 94
  Anti-PRN | 151.4 [127.5 to 179.6] | 209.8 [168.5 to 261.3]

3. Primary Outcome: Anti-Polio Virus Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Month 1, one month after the booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 159 | 81
Titers
  Anti-Polio 1: number analyzed (Participants) | 157 | 75
  Anti-Polio 1 | 2183.3 [1812.4 to 2630.1] | 1876.1 [1472.8 to 2389.7]
  Anti-Polio 2: number analyzed (Participants) | 124 | 71
  Anti-Polio 2 | 2693.1 [2176.3 to 3332.5] | 2203.8 [1681 to 2889.4]
  Anti-Polio 3 | 3762.4 [3080.9 to 4594.6] | 4185.1 [3318.3 to 5278.3]
Statistical Analysis 1: Comparison: Boostrix Polio Group vs Repevax Group; Immune response difference to anti-Polio 1 antigen; Test type: Non-Inferiority — Criterion for evaluation of the corresponding objective: Upper limit (UL) of the 95% confidence interval (CI) on the GMT ratio for the groups' (Repevax Group divided by Boostrix-Polio Group) was lower than or equal to (≤) 2; ANCOVA; Difference in adjusted GMT ratio = 0.91, 95% CI 2-sided [0.65 to 1.28]
Statistical Analysis 2: Comparison: Boostrix Polio Group vs Repevax Group; Immune response difference to anti-Polio 2 antigen; Test type: Non-Inferiority — Criterion for evaluation of the corresponding objective: UL of the 95% CI on the GMT ratio for the groups' (Repevax Group divided by Boostrix-Polio Group) ≤ 2; ANCOVA; Difference in adjusted GMT ratio = 0.78, 95% CI 2-sided [0.54 to 1.12]
Statistical Analysis 3: Comparison: Boostrix Polio Group vs Repevax Group; Immune response difference to anti-Polio 3 antigen; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; ANCOVA; Difference in adjusted GMT ratio = 1.3, 95% CI 2-sided [0.93 to 1.84]

4. Secondary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T)
Description: A seroprotected subject was defined a subject with anti-D and anti-T antibody concentrations ≥ 0.1 international units per millilitre (IU/mL).
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 195 | 96
Participants
  Anti-D, M0: number analyzed (Participants) | 177 | 90
  Anti-D, M0 | 136 | 75
  Anti-D, M1 | 195 | 96
  Anti-T, M0: number analyzed (Participants) | 177 | 90
  Anti-T, M0 | 116 | 63
  Anti-T, M1: number analyzed (Participants) | 194 | 96
  Anti-T, M1 | 194 | 96

5. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN
Description: A seropositive subject for anti-PT, anti-FHA and anti-PRN was a subject whose antibody concentration was ≥ 5 EL.U/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 195 | 96
Participants
  Anti-PT, M0: number analyzed (Participants) | 171 | 90
  Anti-PT, M0 | 31 | 18
  Anti-PT, M1: number analyzed (Participants) | 194 | 96
  Anti-PT, M1 | 194 | 96
  Anti-FHA, M0: number analyzed (Participants) | 174 | 85
  Anti-FHA, M0 | 112 | 60
  Anti-FHA, M1: number analyzed (Participants) | 195 | 95
  Anti-FHA, M1 | 195 | 95
  Anti-PRN, M0: number analyzed (Participants) | 175 | 91
  Anti-PRN, M0 | 61 | 37
  Anti-PRN, M1: number analyzed (Participants) | 195 | 94
  Anti-PRN, M1 | 194 | 94

6. Secondary Outcome: Number of Seroprotected Subjects Against Polio Type 1, 2 and 3
Description: A seroprotected subject was defined as a subject with anti-polio type 1, 2 and 3 antibody titres ≥ the value of 8.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 160 | 81
Participants
  Anti-polio 1, M0: number analyzed (Participants) | 160 | 77
  Anti-polio 1, M0 | 95 | 49
  Anti-polio 1, M1: number analyzed (Participants) | 157 | 75
  Anti-polio 1, M1 | 156 | 75
  Anti-polio 2, M0: number analyzed (Participants) | 159 | 79
  Anti-polio 2, M0 | 109 | 55
  Anti-polio 2, M1: number analyzed (Participants) | 124 | 71
  Anti-polio 2, M1 | 123 | 71
  Anti-polio 3, M0: number analyzed (Participants) | 156 | 79
  Anti-polio 3, M0 | 100 | 47
  Anti-polio 3, M1: number analyzed (Participants) | 159 | 81
  Anti-polio 3, M1 | 158 | 81

7. Secondary Outcome: Number of Seropositive Subjects for Anti-measles Antibody
Description: A seropositive subject was defined as a subject with anti-measles antibody titers ≥ 150 mIU/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 159 | 76
Participants
  Anti-Measles, M0 | 155 | 74
  Anti-Measles, M1: number analyzed (Participants) | 136 | 68
  Anti-Measles, M1 | 136 | 68

8. Secondary Outcome: Number of Seropositive Subjects for Anti-mumps Antibody
Description: A seropositive subject was defined as a subject with anti-mumps antibody titers ≥ 231 U/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 156 | 76
Participants
  Anti-Mumps, M0 | 140 | 69
  Anti-Mumps, M1: number analyzed (Participants) | 133 | 68
  Anti-Mumps, M1 | 133 | 68

9. Secondary Outcome: Number of Seropositive Subjects for Anti-rubella Antibody
Description: A seropositive subject was defined as a subject with anti-rubella antibody titers ≥ 4 IU/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 158 | 76
Participants
  Anti-Rubella, M0 | 158 | 76
  Anti-Rubella, M1: number analyzed (Participants) | 134 | 68
  Anti-Rubella, M1 | 134 | 68

10. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in IU/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 195 | 96
IU/mL
  Anti-D, M0: number analyzed (Participants) | 177 | 90
  Anti-D, M0 | 0.228 [0.194 to 0.267] | 0.259 [0.209 to 0.32]
  Anti-D, M1 | 8.113 [7.259 to 9.068] | 11.948 [10.003 to 14.271]
  Anti-T, M0: number analyzed (Participants) | 177 | 90
  Anti-T, M0 | 0.209 [0.173 to 0.253] | 0.241 [0.184 to 0.315]
  Anti-T, M1: number analyzed (Participants) | 194 | 96
  Anti-T, M1 | 6.787 [5.961 to 7.727] | 9.194 [7.565 to 11.175]

11. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: At Month 0, before the booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 175 | 91
EL.U/mL
  Anti-PT: number analyzed (Participants) | 171 | 90
  Anti-PT | 3.4 [3 to 3.9] | 3.2 [2.9 to 3.6]
  Anti-FHA: number analyzed (Participants) | 174 | 85
  Anti-FHA | 12.9 [10 to 16.6] | 10.7 [7.9 to 14.5]
  Anti-PRN | 4.3 [3.8 to 5] | 4.3 [3.7 to 5]

12. Secondary Outcome: Anti-mumps Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in U/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 156 | 76
U/mL
  Anti-Mumps, M0 | 1035.3 [869.8 to 1232.3] | 971.7 [752.1 to 1255.5]
  Anti-Mumps, M1: number analyzed (Participants) | 133 | 68
  Anti-Mumps, M1 | 6801.9 [6155 to 7516.8] | 6219.4 [5365.8 to 7208.8]

13. Secondary Outcome: Anti-measles Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in mIU/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 159 | 76
mIU/mL
  Anti-Measles, M0 | 2644 [2261.3 to 3091.6] | 2702.6 [2146 to 3403.6]
  Anti-Measles, M1: number analyzed (Participants) | 136 | 68
  Anti-Measles, M1 | 3817.7 [3422.3 to 4258.8] | 3798 [3262.6 to 4421.1]

14. Secondary Outcome: Anti-rubella Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in IU/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 158 | 76
IU/mL
  Anti-Rubella, M0 | 66.5 [59.1 to 74.8] | 72.6 [59.8 to 88.1]
  Anti-Rubella, M1: number analyzed (Participants) | 134 | 68
  Anti-Rubella, M1 | 134.3 [120.7 to 149.4] | 130.3 [111.7 to 152]

15. Secondary Outcome: Anti-Polio Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Month 0, before the booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 160 | 79
Titers
  Anti-Polio 1: number analyzed (Participants) | 160 | 77
  Anti-Polio 1 | 12.8 [10.6 to 15.5] | 13.2 [10.2 to 17.1]
  Anti-Polio 2: number analyzed (Participants) | 159 | 79
  Anti-Polio 2 | 15.5 [12.8 to 18.8] | 14.6 [11.3 to 18.8]
  Anti-Polio 3: number analyzed (Participants) | 156 | 79
  Anti-Polio 3 | 15.4 [12.7 to 18.8] | 14.5 [10.4 to 20.1]

16. Secondary Outcome: Number of Subjects With a Booster Response to PT, FHA and PRN Antigens
Description: Booster response was defined as: For initially seronegative subjects (pre-vaccination concentration < 5 EL.U/mL), antibody concentrations at least four times the assay cut-off (post vaccination concentration ≥ 20 EL.U/mL). For initially seropositive subjects (with pre-vaccination concentration ≥ 5 EL.U/mL and < 20 EL.U/mL), an increase in antibody concentrations of at least four times the Pre booster vaccination concentration. For initially seropositive subjects (with pre-vaccination concentration ≥ 20 EL.U/mL), an increase in antibody concentrations of at least two times the Pre booster vaccination concentration.
Time Frame: At Month 1, one month after the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 175 | 90
Participants
  Anti-PT: number analyzed (Participants) | 170 | 90
  Anti-PT | 154 | 73
  Anti-FHA: number analyzed (Participants) | 174 | 85
  Anti-FHA | 165 | 79
  Anti-PRN: number analyzed (Participants) | 175 | 89
  Anti-PRN | 169 | 89

17. Secondary Outcome: Number of Subjects With Booster Response for Polio Type 1, 2 and 3 Antigens
Description: Booster response defined as: For initially seronegative subjects, antibody titers at least four times the cut-off (post-vaccination titer ≥ 32); For initially seropositive subjects, an increase in antibody titers of at least four times the Pre booster vaccination titer.
Time Frame: At Month 1, one month after the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 131 | 68
Participants
  Anti-Polio 1: number analyzed (Participants) | 131 | 63
  Anti-Polio 1 | 129 | 63
  Anti-Polio 2: number analyzed (Participants) | 100 | 61
  Anti-Polio 2 | 99 | 59
  Anti-Polio 3: number analyzed (Participants) | 126 | 68
  Anti-Polio 3 | 124 | 68

18. Secondary Outcome: Number of Seroconverted Subjects for Anti-measles
Description: Seroconversion for anti-measles was defined as the appearance of antibodies after vaccination in subjects who were initially seronegative [with antibody concentrations ≥ 150 milli-international units per millilitre (mIU/mL)].
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 4 | 2
Participants
  Anti-measles, M0 | 0 | 0
  Anti-measles, M1 | 4 | 2

19. Secondary Outcome: Number of Seroconverted Subjects for Anti-mumps
Description: Seroconversion for anti-mumps was defined as the appearance of antibodies after vaccination in subjects who were initially seronegative [with antibody concentrations ≥ 231 units per millilitre (U/mL)].
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 16 | 7
Participants
  Anti-mumps, M0 | 0 | 0
  Anti-mumps, M1: number analyzed (Participants) | 11 | 6
  Anti-mumps, M1 | 11 | 6

20. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented, who had their symptoms sheet filled in and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 255 | 125
Participants
  Any Pain | 127 | 70
  Any Redness | 146 | 73
  Any Swelling | 92 | 53

21. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 255 | 125
Participants
  Any Drowsiness | 77 | 39
  Any Irritability | 107 | 49
  Any Loss of appetite | 67 | 30
  Any Temperature | 18 | 9

22. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 255 | 130
Participants | 88 | 36

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (From Day 0 to Month 1)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Repevax Group
Number analyzed (Participants) | 255 | 130
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) following vaccination. Unsolicited adverse events: during the 31-day (Days 0-30) following vaccination. Serious adverse events: during the entire study period (from Month 0 to Month 1).
Arm/Group | Boostrix Polio Group | Repevax Group
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/130
Serious Adverse Events (participants affected / at risk) | 1/255 | 0/130
Other Adverse Events (participants affected / at risk) | 215/255 | 108/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Polio Group (N=255) | Repevax Group (N=130)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Polio Group (N=255) | Repevax Group (N=130)
Pain (General disorders) | 127 | 70 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (General disorders) | 146 | 73 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (General disorders) | 92 | 53 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (General disorders) | 77 | 39 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Irritability (General disorders) | 107 | 49 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (General disorders) | 67 | 30 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Temperature (Axillary) (General disorders) | 18 | 9 — This solicited general symptom was only collected from subjects with their symptom sheets completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.